CLINICAL TRIAL: NCT05174910
Title: Investigation of the Benefit of Using an Autologous Platelet-rich Fibrin Matrix (Obsidian ASG®) for Treatment of Anastomosis During Rectal Surgery - a Single-blind, Randomized, Multicenter Pilot Study
Brief Title: Investigation of the Benefit of Using an Autologous Platelet-rich Fibrin Matrix (Obsidian ASG®) for Treatment of Anastomosis During Rectal Surgery
Acronym: ORSY
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vivostat (Industry)
Collaborators: Raffeiner GmbH (Industry); European Commission (Other); AF Schimetta GMbH (Unknown); Rivolution GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ORSY
Record Dates: First submitted 2021-11-30; First posted 2022-01-03 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Anastomotic Leak Rectum

STUDY DESIGN:
Intervention Model Description: Multicenter, prospective, randomized, single-blind
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With Obsidian ASG (Active Comparator): Anastomosis treatment using standard procedure and Obsidian ASG
  Interventions: Device: Obsidian ASG
- Without Obsidian ASG (No Intervention): Anastomosis treatment using standard procedure

INTERVENTIONS:
Device: Obsidian ASG — Application of an autologous platelet-rich fibrin matrix
  Arms: With Obsidian ASG

SUMMARY:
Anastomotic insufficiency remains one of the most significant problems after rectal resection.The complications following anastomotic insufficiency leads to increased morbidity and mortality with subsequent prolongation of hospital stay and higher costs.

This study is an investigation of the benefit of using an autologous platelet-rich fibrin matrix (Obsidian ASG®) for treatment of anastomosis during rectal surgery - a single-blind, randomized, multicenter pilot study with enrollment of 2x125 patients

The main objective of the study is to investigate on an exploratory basis whether the use of Obsidian ASG® during rectal resection reduces the frequency of postoperative anastomotic insufficiency compared to standard anastomotic technique.

The secondary objectives of the study are to investigate on an exploratory basis:

* The frequency of anastomotic insufficiency (ISREC Criteria) severity
* Staple line bleeding requiring surgical intervention
* The duration of postoperative hospitalization are reduced when using Obsidian ASG ® compared with standard anastomotic treatment alone.

are reduced when Obsidian ASG ® is added to the standard of anastomotic treatment compared with standard anastomotic treatment alone.

ELIGIBILITY:
Inclusion Criteria:

The following inclusion criteria will be considered:

* Written informed consent
* Age > 18 years
* Indication for elective oncological rectal resection in the presence of malignant rectal disease and the lower edge of the tumor, measured from the anal verge with the rigid rectoscope, ≤ 14cm
* Use of a circular anastomosis using the "double stapling technique"(6) during creation of the anastomosis
* Expected availability within the maximum 45-day period of study participation
* The use of "golden standard" stapling technology devices; 3 rows endo linear stapler; 2 rows circular stapling devices should be used in an open and laparoscopic approach

Exclusion Criteria:

The following exclusion criteria will be considered:

* Pregnancy, or the non-exclusion of pregnancy (for women of childbearing potential). In the case of menopause having occurred more than 2 years ago or postmenopausal sterilization or surgical sterilization, the authorized physician is free to classify the female study participant as non-pregnant, so that the pregnancy test otherwise required at the beginning of study participation (or during subject screening) may be omitted.
* Risk of pregnancy occurring while taking part in the study in women not meeting at least one of the following criteria: Onset of menopause more than 2 years ago, postmenopausal sterilization, surgical sterilization, a promise to use contraception (with hormones, coil or diaphragm/condom + spermicide), while enrolled in the study) In the case of onset of menopause more than 2 years ago, postmenopausal sterilization or surgical sterilization, the authorized doctor is free to classify the patient in question as infertile. Furthermore, it is at the discretion of the authorized physician to classify the patient in question on the basis of continuous inpatient care in such a way that the occurrence of pregnancy during participation in the study can be ruled out ("continuous determination of the absence of pregnancy"). If one of the above classifications applies, further measures to ensure that a pregnancy does not occur during the patient's participation in the study may not be required.
* Breastfeeding period
* Lack of legal capacity
* Vulnerable persons according to the law
* Comorbidity with the potential for relevant impairment of anastomosis durability (leukemia, cirrhosis of the liver, Child Pugh C, etc.)
* Preoperative anemia with Hb <8g/dL
* Participating in another study
* Patients on Aspirin not able to stop using Aspirin for medical reasons minimum 3 days before taking the blood sampling.
* Patients on Clopidogrel not able to stop using Clopidogrel for medical reasons minimum 7 days before blood sampling.
* Patients on other platelet aggregation inhibitor therapies
* Contraindication for Obsidian ASG®
* Surgical technique of transanal total mesorectal excision (TaTME)
* Application of a circular powered stapler in the course of anastomosis supply with GSTTM technology or a 3 row circular stapler use while creating the study anastomosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-12-23 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Anastomosis insufficiency [yes/no] | 45 days
  Anastomosis insufficiency after colorectal surgery with primary anastomosis

SECONDARY OUTCOMES:
Anastomotic insufficiency [0/A/B/C]* | 45 days
  *ISREC, International Study Group of Rectal Cancer - severity grading of anastomotic leakage
Staple suture line bleeding requiring surgical intervention [yes, with surgical intervention / yes, without surgical intervention / no] | 45 days
  Staple suture line bleeding requiring surgical intervention
Postoperative hospital length of stay [days] | 45 days
  Days spent in hospital after undergoing colorectal surgery

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Shamiyeh, Prim.Doz.Dr., Principal Investigator — Kepler Universitätsklinikum Gmbh
Locations (13):
- Austria (4):
  - Krankenhaus der Barmherzigen Brûder, Graz
  - Kepler Universitätsklinikum GmbH, Med campus III, Linz
  - Krankenhaus der Barmherzigen Brüder Wien, Vienna
  - Landesklinikum Wienerneustadt, Wiener Neustadt
- Germany (5):
  - RoMed Klinikum Rosenheim, Rosenheim, Bavaria
  - Universität Augsburg, Augsburg
  - Diakonissenkrankenhaus Dresden, Dresden
  - Klinikum Fürth, Fürth
  - Klinikum Nürnberg Nord, Nuremberg
- University Milano, Milan, Italy
- University Hospital Belgrade, Belgrade, Serbia
- Spain (2):
  - Granada Hospital, Granada
  - Consorci Hospital General Universitari de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No